CLINICAL TRIAL: NCT04891796
Title: Tobacco Control Policy-related Survey by Landline and Mobile Telephone
Brief Title: Tobacco Control Policy-related Survey 2020
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Associate Professor, The University of Hong Kong
Other Study IDs: 2020 Policy Survey
Record Dates: First submitted 2021-05-17; First posted 2021-05-18 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Survey on Tobacco Control
Keywords: Smoking; Tobacco Control Policy; Tobacco Control Measures
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Current smokers: Individuals who, at the time of the survey, smoke any forms of tobacco product either daily or occasionally.
  Interventions: Other: No intervention
- Ex-smokers: Individuals who were formerly smokers but, at the time of the survey, do not smoke at all.
  Interventions: Other: No intervention
- Never Smokers: Individuals who, at the time of the survey, have never smoked at all.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Aim: to collect further information on issues related to tobacco control which should be addressed and advocated in further tobacco control measures in Hong Kong

The objectives of this policy-related survey by landline and mobile telephone are as follows:

1. to update information on prevalence of conventional cigarettes, e-cigarettes, heat-not-burn tobacco products and waterpipe tobaccos ;
2. to investigate the effects of new pictorial health warning policy in the public;
3. to investigate the level of public support on current and future tobacco control measures and taxation;
4. to address the timely impacts of smoke-free policies, public support for further tobacco control measures and assist COSH in shaping policy direction for government;

Current study is a cross-sectional retrospective landline and mobile telephone survey based on questionnaires. The target sample size is planned to be 5,100 Hong Kong residents, including 1,700 current, ex and never smokers respectively. All three smoking status are to be evenly sampled by landline and mobile telephone. All data will be collected using a Computer Assisted Telephone Interview (CATI) system, which allows real-time data capture and consolidation. All interviews shall be conducted anonymously except for those who are willing to participate subsequent studies pictorial warning opinion. Analysis of survey data will aim to identify current opinion on tobacco control policies and implications for future policies. All eligible subjects who complete the telephone survey will be included in the analysis. Comparison with past trends conducted by previous landline and mobile phone surveys and, where possible, extrapolation of future trends will be explored. Weightings will be applied to adjust for the sex and age of Hong Kong population, and to handle the over-sampling issues of ex- and current smokers. The data analysis will be conducted by experienced statisticians in the applicants' team.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong resident aged 15 and above
* Cantonese speakers

Exclusion Criteria:

* Unable to provide a consent
* Speak language other than Cantonese

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Hong Kong residents
Sampling Method: Probability Sample
Enrollment: 5112 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
Attitudes toward tobacco control policies | Finish all telephone interviews by Sep 2021
  Topic includes cigarette consumption and dependence, heat-not-burn tobacco products, e-cigarettes, waterpipe tobaccos, years of abstinence, intention to quit, influence of COVID-19 on smoking behaviour, tobacco endgame, second-hand smoke exposure, pictorial health warning, smoke-free areas, tobacco tax increase, peer influence on smoking, and current use and acceptance of phone-based intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The Hong Kong Public Opinion Research Institute, Hong Kong, Hong Kong